CLINICAL TRIAL: NCT00134381
Title: The Effects of Topically Applied Constituents of Green Tea on UV Induced Increase in p53 and Apoptotic Markers in the Skin of Human Volunteers
Brief Title: Green Tea and Ultraviolet Light-induced Skin Damage
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator left institution before study could complete.
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3808
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Normal volunteer study
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active drug (Active Comparator): bilateral comparison of green tea constituent
  Interventions: Drug: Green Tea
- placebo (Placebo Comparator): bilateral comparison of placebo vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Green Tea — Green tea product (EGCG or caffeine) in vehicle will be applied immediately after and at sequential time points after exposure of a 5x5-cm area of skin to a dose of UVB that is 0.5-2 times the subject's minimal erythema dose (MED)
  Arms: active drug
Drug: Placebo — Placebo (vehicle alone) will be applied immediately after and at sequential time points after exposure of a 5x5-cm area of skin to a dose of UVB that is 0.5-2 times the subject's minimal erythema dose (MED)
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate whether topically applied constituents of green tea [caffeine or (-)-epigallocatechin gallate; EGCG] have a protective effect on skin exposed to ultraviolet light (UV).

DETAILED DESCRIPTION:
The purpose of this study is to investigate if topically applied constituents of green tea [caffeine or (-) - epigallocatechin gallate; EGCG] have a protective effect on skin exposed to ultraviolet light (UV). In the double-blinded study all subjects will receive 311 nanometer UVB light at a dose that is 0.5-1.5X their individual minimal erythema dose (MED). One part of the experiment will involve applying a topical natural product (caffeine or EGCG) and placebo to bilateral symmetric sites. The natural product and the placebo will be applied immediately after and at 1/2 hour, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 24 hours, 25 hours, and 27 hours after exposure to a 0.5-1.5 MED dose of UV light. Another part of the study involves performing skin biopsies. One will be done prior to UVB exposure, 2 will be done at 24 hours and 2 more will be done at 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be normal adult volunteers who are 18 to 65 years of age.

Exclusion Criteria:

* Subjects who drink more than two cups of coffee, tea, or caffeinated soda/beverages per day.
* Subjects who are unable to get an erythemic response (i.e., a sunburn).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2003-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Magliocco, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ Division of Clinical Pharmacology, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- EGCG in Acetone Vehicle (L Side: Active; R Side: Placebo): bilateral comparison Subjects randomized to this group received applications of EGCG to a test site on the left side of the body and placebo to a test site on the right side of the body.
- EGCG in Acetone Vehicle (R Side: Active; L Side: Placebo): bilateral comparison Subjects randomized to this group received applications of EGCG to a test site on the right side of the body and placebo to a test site on the left side of the body.
- Caffeine in Acetone Vehicle (L Side: Active; R Side: Placebo); Caffeine in Cream Vehicle (L Side: Active; R Side: Placebo): bilateral comparison Subjects randomized to this group received applications of caffeine to a test site on the left side of the body and placebo to a test site on the right side of the body.
- Caffeine in Acetone Vehicle (R Side: Active; L Side: Placebo); Caffeine in Cream Vehicle (R Side: Active; L Side: Placebo): bilateral comparison Subjects randomized to this group received applications of caffeine to a test site on the right side of the body and placebo to a test site on the left side of the body.
Period: Overall Study
Arm/Group | EGCG in Acetone Vehicle (L Side: Active; R Side: Placebo) | EGCG in Acetone Vehicle (R Side: Active; L Side: Placebo) | Caffeine in Acetone Vehicle (L Side: Active; R Side: Placebo) | Caffeine in Acetone Vehicle (R Side: Active; L Side: Placebo) | Caffeine in Cream Vehicle (L Side: Active; R Side: Placebo) | Caffeine in Cream Vehicle (R Side: Active; L Side: Placebo)
Started | 1 | 2 | 1 | 2 | 31 | 31
Completed | 1 | 2 | 1 | 2 | 31 | 29
Not Completed | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Bilateral Comparison: In this bilateral comparison study, subjects were randomized to receive applications of green tea product or placebo to test sites on the left and right sides of the body.
Arm/Group | Bilateral Comparison
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 66
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Change in UVB-Induced Active Caspase-3-Positive Keratinocytes by Green Tea Compounds
Description: The mean change in number of active caspase-3+ apoptotic keratinocytes between 0- and 48-hour time points was calculated for skin biopsy samples of subjects who had been exposed to UVB on symmetrical right and left test sites which were then randomized to receive active test substance (EGCG or caffeine) or placebo (vehicle) at sequential time points after UVB exposure.
Time Frame: 48 hrs
Population: Six (6) subjects were randomized (split-body) to receive either EGCG (3 subjects) or caffeine (3 subjects) in acetone vehicle on a test site on one side of the body and placebo (acetone vehicle) on the test site on the other side of the body, after exposure to twice the individual subjects' minimal erythema dose (MED) of UVB.
Measure: Mean (Standard Error); unit: cells/mm
Groups:
- EGCG in Acetone Vehicle: bilateral comparison Subjects were randomized to receive applications of EGCG (28.3 mg/mL; active drug) on the test site on one side of the body after exposure to UVB that was twice their individual minimal erythema dose (MED).
- Placebo (Acetone Vehicle in Subjects Who Received EGCG); Placebo (Acetone Vehicle in Subjects Who Received Caffeine): bilateral comparison Subjects were randomized to receive applications of acetone vehicle (placebo) on the test site on one side of the body after exposure to UVB that was twice their individual minimal erythema dose (MED).
- Caffeine in Acetone Vehicle: bilateral comparison Subjects were randomized to receive applications of caffeine (12 mg/mL; active drug) on the test site on one side of the body after exposure to UVB that was twice their individual minimal erythema dose (MED).
Arm/Group | EGCG in Acetone Vehicle | Placebo (Acetone Vehicle in Subjects Who Received EGCG) | Caffeine in Acetone Vehicle | Placebo (Acetone Vehicle in Subjects Who Received Caffeine)
Number analyzed (Participants) | 3 | 3 | 3 | 3
cells/mm | 28.34 (18.51) | 13.05 (9.98) | 10.68 (3.61) | 32.60 (28.14)

2. Primary Outcome: Change in UVB-Induced Apoptotic "Sunburn" Cells by Green Tea Compounds
Description: The mean change in number of apoptotic "sunburn" cells between 0- and 48-hour time points was calculated for skin biopsy samples of subjects who had been exposed to UVB on symmetrical right and left test sites which were then randomized to receive active test substance (EGCG or caffeine) or placebo (vehicle) at sequential time points after UVB exposure.
Time Frame: 48 hr
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cells/mm
Arm/Group | EGCG in Acetone Vehicle | Placebo (Acetone Vehicle in Subjects Who Received EGCG) | Caffeine in Acetone Vehicle | Placebo (Acetone Vehicle in Subjects Who Received Caffeine)
Number analyzed (Participants) | 3 | 3 | 3 | 3
cells/mm | 18.94 (8.18) | 14.79 (7.43) | 28.86 (8.00) | 43.62 (29.22)

3. Primary Outcome: Effect of Topical Applications of 4-6% Caffeine on UVB-Induced Increases in Apoptotic "Sunburn" Cells
Description: The percentage of apoptotic "sunburn" cells was identified in the 48-hr time point skin biopsy samples of subjects who had been exposed to UVB on symmetrical right and left test sites which were then randomized to receive 4-6% caffeine in cream vehicle or placebo (cream vehicle) at sequential time points after UVB exposure.
Time Frame: 48 hr
Population: Twenty (20) subjects received caffeine on one test site and placebo on the other site after exposure to individual subjects' minimal erythema dose (MED) of UVB.Twenty-six (26) subjects received caffeine on one test site and placebo on the other site after exposure to UVB that was 1.5 times subjects' individual minimal erythema dose (MED).
Measure: Mean (Standard Error); unit: percentage of "sunburn" cells
Groups:
- Caffeine in Vehicle Cream (1.0 MED Group): bilateral comparison Subjects were randomized to receive applications of 6% caffeine (active drug) on the test site on one side of the body after exposure to UVB at the subjects' individual minimal erythema dose (MED).
- Placebo Cream (1.0 MED Group): bilateral comparison Subjects were randomized to receive applications of cream vehicle (placebo) on the test site on one side of the body after exposure to UVB at the subjects' individual minimal erythema dose (MED).
- Caffeine in Vehicle Cream (1.5 MED Group): bilateral comparison Subjects were randomized to receive applications of 4-6% caffeine (active drug) on the test site on one side of the body after exposure to UVB that was 1.5 times subjects' individual minimal erythema dose (MED).
- Placebo Cream (1.5 MED Group): bilateral comparison Subjects were randomized to receive applications of cream vehicle (placebo) on the test site on one side of the body after exposure to UVB that was 1.5 times subjects' individual minimal erythema dose (MED).
Arm/Group | Caffeine in Vehicle Cream (1.0 MED Group) | Placebo Cream (1.0 MED Group) | Caffeine in Vehicle Cream (1.5 MED Group) | Placebo Cream (1.5 MED Group)
Number analyzed (Participants) | 20 | 20 | 26 | 26
percentage of "sunburn" cells | 7.50 (2.06) | 4.93 (1.54) | 5.10 (0.80) | 4.63 (0.60)

4. Primary Outcome: Effect of Topical Applications of 4-6% Caffeine on UVB-Induced Increases in Caspase-3-Positive Cells
Description: The percentage of caspase-3-positive cells was identified in the 48-hr time point skin biopsy samples of subjects who had been exposed to UVB on symmetrical right and left test sites which were then randomized to receive 4-6% caffeine in cream vehicle or placebo (cream vehicle) at sequential time points after UVB exposure.
Time Frame: 48 hr
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percentage of caspase-3-positive cells
Arm/Group | Caffeine in Vehicle Cream (1.0 MED Group) | Placebo Cream (1.0 MED Group) | Caffeine in Vehicle Cream (1.5 MED Group) | Placebo Cream (1.5 MED Group)
Number analyzed (Participants) | 20 | 20 | 26 | 26
percentage of caspase-3-positive cells | 6.54 (1.85) | 4.53 (1.16) | 4.38 (0.92) | 3.15 (0.46)

5. Primary Outcome: Effect of Topical Applications of 4-6% Caffeine on UVB-Induced Increases in Phospho-p53 (Ser15) Positive Cells
Description: The percentage of phospho-p53 (Ser15) positive cells was identified in the 48-hr time point skin biopsy samples of subjects who had been exposed to UVB on symmetrical right and left test sites which were then randomized to receive 4-6% caffeine in cream vehicle or placebo (cream vehicle) at sequential time points after UVB exposure.
Time Frame: 48 hr
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percentage of p-p53 (Ser15) pos. cells
Arm/Group | Caffeine in Vehicle Cream (1.0 MED Group) | Placebo Cream (1.0 MED Group) | Caffeine in Vehicle Cream (1.5 MED Group) | Placebo Cream (1.5 MED Group)
Number analyzed (Participants) | 20 | 20 | 26 | 26
percentage of p-p53 (Ser15) pos. cells | 13.03 (2.40) | 13.46 (2.47) | 15.98 (2.17) | 15.15 (2.57)

6. Secondary Outcome: Effect of Green Tea Compounds on UVB-Induced Erythema
Description: Erythema of the right and left test sites was scored on a scale of 0-3 (0 = no evidence [no erythema]; 1 = mild [pink or light red color]; 2 = moderate [red color]; 3 = severe [very red or dark color]) including half-integer grading. Scoring was performed immediately after UVB exposure and at sequential time points thereafter. The mean scores at 48 hr were calculated.
Time Frame: 48 hrs
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | EGCG in Acetone Vehicle | Placebo (Acetone Vehicle in Subjects Who Received EGCG) | Caffeine in Acetone Vehicle | Placebo (Acetone Vehicle in Subjects Who Received Caffeine)
Number analyzed (Participants) | 3 | 3 | 3 | 3
units on a scale | 1.33 (0.44) | 1 (0) | 1.17 (0.17) | 1.33 (0.44)

7. Secondary Outcome: Effect of 4-6% Caffeine on UVB-Induced Erythema
Description: Erythema of the right and left test sites was scored on a scale of 0-3 (0 = no evidence [no erythema]; 1 = mild [pink or light red color]; 2 = moderate [red color]; 3 = severe [very red or dark color]) including half-integer grading. Scoring was performed immediately after UVB exposure and at sequential time points thereafter. The erythema scores at 6, 8, and 24 hr post-UVB were averaged.
Time Frame: 24 hr
Population: Sixty-two (62) subjects received caffeine on one test site and placebo on the other site after exposure to 0.5-1.5 times individual subjects' minimal erythema dose (MED) of UVB.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Caffeine in Vehicle Cream (0.5 MED Group): bilateral comparison Subjects were randomized to receive applications of 6% caffeine (active drug) on the test site on one side of the body after exposure to UVB at 0.5 times the subjects' individual minimal erythema dose (MED).
- Placebo Cream (0.5 MED Group): bilateral comparison Subjects were randomized to receive applications of cream vehicle (placebo) on the test site on one side of the body after exposure to UVB at 0.5 times the subjects' individual minimal erythema dose (MED).
Arm/Group | Caffeine in Vehicle Cream (0.5 MED Group) | Placebo Cream (0.5 MED Group) | Caffeine in Vehicle Cream (1.0 MED Group) | Placebo Cream (1.0 MED Group) | Caffeine in Vehicle Cream (1.5 MED Group) | Placebo Cream (1.5 MED Group)
Number analyzed (Participants) | 12 | 12 | 21 | 21 | 29 | 29
units on a scale | 0.18 (0.04) | 0.38 (0.05) | 0.66 (0.06) | 0.83 (0.05) | 1.14 (0.05) | 1.36 (0.05)

ADVERSE EVENTS:
Groups:
- Bilateral Comparison: In this bilateral comparison study, subjects were randomized to receive applications of green tea product or placebo to test sites on the left and right sides of the body after exposure of the test sites to UVB.
Arm/Group | Bilateral Comparison
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 6/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral Comparison (N=68)
menstrual cramps (Reproductive system and breast disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
tenderness of right test site (Skin and subcutaneous tissue disorders) | 1 (1)
superficial wound infection (Infections and infestations) | 1 (1)
headache (Nervous system disorders) | 1 (1)
tooth abscess (Infections and infestations) | 1 (1)
accidental removal of a suture (Skin and subcutaneous tissue disorders) | 1 (1)
rash over adhesive area (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No